CLINICAL TRIAL: NCT03630497
Title: A Randomised, Double-blind, Placebo-controlled, Single (SAD) and Multiple Ascending Dose (MAD) Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BN201 in Healthy Subjects
Brief Title: BN201 SAD MAD Study in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Accure Therapeutics (Industry)
Collaborators: Simbec Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BN201_RDREG_251; 2017-001202-14 (EudraCT Number)
Record Dates: First submitted 2018-07-23; First posted 2018-08-15 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Optic Neuritis; Optic; Neuritis, With Demyelination
Keywords: Acute Optic Neuritis (AON); Demyelination; Optic Neuritis
MeSH Terms: conditions — Optic Neuritis; Neuritis; Demyelinating Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Period 1 Single Dose SD1 (first dose) (Experimental): Period 1 Group SD1 a single IV infusion of first single dose of BN201 (n=6) or placebo (n=2)
  Comparison of BN201 treatment with Placebo
  Interventions: Drug: Comparison of BN201 treatment with Placebo
- Period 1 Single Dose SD2 (second dose) (Experimental): Period 1 Group SD2 a single IV infusion of second single dose of BN201 (n=6) or placebo (n=2)
  Comparison of BN201 treatment with Placebo
  Interventions: Drug: Comparison of BN201 treatment with Placebo
- Period 1 Single Dose SD3 (third dose) (Experimental): Period 1 Group SD3 a single IV infusion of third single dose of BN201 (n=6) or placebo (n=2)
  Comparison of BN201 treatment with Placebo
  Interventions: Drug: Comparison of BN201 treatment with Placebo
- Period 1 Single Dose SD4 (fourth dose) (Experimental): Period 1 Group SD4 a single IV infusion of fourth single dose of BN201 (n=6) or placebo (n=2)
  Comparison of BN201 treatment with Placebo
  Interventions: Drug: Comparison of BN201 treatment with Placebo
- Period 2 Single Dose SD1 (fifth dose) (Experimental): Period 2 Group SD1 a single IV infusion of fifth single dose of BN201 (n=6) or placebo (n=2)
  Comparison of BN201 treatment with Placebo
  Interventions: Drug: Comparison of BN201 treatment with Placebo
- Period 2 Single Dose SD2 (sixth dose) (Experimental): Period 2 Group SD2 a single IV infusion of sixth single dose of BN201 (n=6) or placebo (n=2)
  Comparison of BN201 treatment with Placebo
  Interventions: Drug: Comparison of BN201 treatment with Placebo
- Period 2 Single Dose SD3 (seventh dose) (Experimental): Period 2 Group SD3 a single IV infusion of seventh single dose of BN201 (n=6) or placebo (n=2)
  Comparison of BN201 treatment with Placebo
  Interventions: Drug: Comparison of BN201 treatment with Placebo
- Period 2 Single Dose SD4 (Optional) (Experimental): (Optional) Period 2 Group SD4 a single IV infusion of eighth single dose of BN201 (n=6) or placebo (n=2)
  Comparison of BN201 treatment with Placebo
  Interventions: Drug: Comparison of BN201 treatment with Placebo
- Multiple Dose MD1 (Experimental): MD1 once daily IV infusions of first multiple dose BN201 (n=6) or placebo (n=2) for 5 consecutive days
  Comparison of BN201 treatment with Placebo
  Interventions: Drug: Comparison of BN201 treatment with Placebo
- Multiple Dose MD2 (Experimental): MD2 once daily IV infusions of second multiple dose BN201 (n=6) or placebo (n=2) for 5 consecutive days
  Comparison of BN201 treatment with Placebo
  Interventions: Drug: Comparison of BN201 treatment with Placebo

INTERVENTIONS:
Drug: Comparison of BN201 treatment with Placebo — Single Dose or Multiple Dose of BN201 IV administration
  Other Names: BN201

SUMMARY:
The purpose of this study is to investigate the safety, tolerability, pharmacokinetics, and pharmacodynamics of single and multiple doses of BN201 in healthy subjects.

This is a phase I, randomised, double-blind, placebo-controlled study to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of BN201 in healthy subjects following single ascending doses and two cohorts of multiple doses. The study will be conducted in two parts (Part A and Part B). Part A (up to 8 single ascending doses (SD)) will be conducted in 32 subjects (4 interlocking cohorts of 8 subjects). Part B (up to 2 multiple ascending doses (MD)) will be conducted in 16 subjects (2 cohorts of 8 subjects). Subjects in Part A will undergo a screening period (Day -28 to Day -2), two in-patient treatment periods compromising 3 overnight stays (from Day -1 to Day 3) with a wash out period of at least 14 days between dose administrations and a follow up visit 12 to 16 days following administration of IMP. Subjects in Part B will undergo a screening period (Day -28 to Day -2), an in-patient treatment period compromising 7 overnight stays (from Day -1 to Day 7) and a follow up visit 12 to 16 days following final administration of Investigational Medicinal Product (IMP).

DETAILED DESCRIPTION:
Screening (Days -28 to -2) Screening assessments will be performed within 28 days of the first dose to ensure the eligibility of participants. Assessments will include medical history, demographics, concomitant medication check, physical examination, body weight, height, BMI, HIV, Hepatitis B and Hepatitis C screen, drugs of abuse and alcohol screen, routine laboratory assessments (biochemistry, haematology and urinalysis), 12-lead ECG, EEG monitoring, brain MRI scan, vital signs (supine systolic and diastolic blood pressure, pulse) and body temperature. Female participants will also be screened for pregnancy and hormone status. A C-SSRS questionnaire will also be performed at screening for Part B only.

Treatment Period

Part A:

Up to four cohorts ((SD1), (SD2), (SD3), (SD4)) of eight subjects will be randomly assigned to receive either two single intravenous doses of BN201, two single intravenous doses of placebo or one single intravenous dose of BN201 and placebo (per treatment period) over two treatment periods (Period 1 and Period 2). Within each cohort, 6 subjects will receive BN201 and 2 subjects will receive placebo. Two "dose leader" subjects will be dosed on the same day, at least 48 h before the remaining subjects in the cohort. Of these two subjects, one will be dosed with BN201 and the other with placebo. The Chief Investigator (or delegate) must confirm it is safe to continue with the dosing of the remainder of the cohort following review of appropriate safety data. The remaining 6 subjects of the cohort (five randomised to active and one to placebo) will then be dosed.

Subjects will be admitted to the clinical unit in the morning of Day -1 and will remain in the unit until the 48 h post dose scheduled assessments and procedures have been performed (Day 3). On Day -1 of each Treatment Period subjects' eligibility will be re-assessed and blood and urine samples will be collected for laboratory safety tests (including drugs of abuse and alcohol screen, biochemistry, haematology, urinalysis and serum pregnancy test). A 12-lead ECG, vital signs (supine systolic and diastolic blood pressure, pulse), body temperature, adverse event and concomitant medication checks will be performed. The intravenous dose of BN201 or placebo will be based on body weight measured on Day -1. An evening snack will be consumed at least 10 hours (h) before (each) dose administration.

After an overnight fast of at least 10 h, dose administration will occur on the morning of Day 1 between 08:00 and 11:00 whilst subjects are in a semi supine position. The subjects will remain in this position until 2 h post-infusion, however other positions are temporarily allowed for scheduled assessment requirements. Fasting will continue until 4 h after start of infusion; a standardised meal will then be administered.

Subjects will be discharged from the clinical unit on Day 3 (48 h post-dose) providing there are no ongoing safety concerns. There will be a wash out period of at least 14 days between dose administrations prior to subjects returning for their treatment 2 scheduled assessments and procedures.

The following assessments will be made during treatment Period 1 and Period 2:

* Safety assessments: Adverse event (AEs) and concomitant medication check, physical examination, laboratory safety assessments (drugs of abuse and alcohol screen, biochemistry, haematology, urinalysis and serum pregnancy test), 12-lead ECG, telemetry, Holter monitoring, EEG monitoring, vital signs (supine systolic and diastolic blood pressure, pulse) and body temperature, infusion site reaction assessment.
* Pharmacokinetics (PK) assessments: Blood sample collection for measurement of BN201 in plasma.
* Pharmacodynamics (PD) assessments: Blood sample collection for measurement of phosphorylation of N-myc downstream-regulated gene 1 (NDGR1) in peripheral blood mononuclear cells (PBMCs).
* Pharmacogenomic assessments: Blood sample will be collected for potential genotyping of deoxyribonucleic acid (DNA) sequence variants to explore potential relationships with PK/PD and or tolerability.

A follow-up visit (including a brain MRI scan) will be conducted 12 to 16 days following each administration of IMP. If all follow-up assessments are satisfactory to the Investigator following Treatment Period 2 the subject will be discharged from the study. If any AEs are ongoing, or any assessments not satisfactory subjects may be recalled to the unit for follow-up assessments until the Investigator is satisfied the subject may be discharged from the study. Subjects will be advised to return or contact the unit at any time if they may be experiencing any adverse effects.

Enrolment of the subsequent cohort will only proceed, if blinded PK and safety data from the previous cohort has been reviewed by the Sponsor and Chief Investigator and is found to be satisfactory.

Part B:

Two cohorts (MD1, MD2) of eight subjects will be randomly assigned to receive either multiple intravenous doses of BN201 or multiple intravenous doses of placebo once daily for five consecutive days (Day 1 to Day 5). Within each cohort, 6 subjects will receive BN201 and 2 subjects will receive placebo. Two "dose leader" subjects will be dosed on the same day, at least 48 h before the remaining subjects in the cohort. Of these two subjects, one will be dosed with BN201 and the other with placebo. The Chief Investigator (or delegate) must confirm it is safe to continue with the dosing of the remainder of the cohort following review of appropriate safety data. The remaining 6 subjects of the cohort (five randomised to active and one to placebo) will then be dosed. The dose levels to be administered will be based on the safety, tolerability and PK results of Part A. Cohort MD1 can only be started if a higher dose level in the SAD part was well tolerated and that simulated PK modelling for multiple dose administration based on PK data from single doses do not suggest that the Cmax threshold of 13.3 μg/mL will be exceeded. Enrolment of MD2 will only proceed if blinded PK and safety data from subjects in MD1 has been reviewed by the Sponsor and Chief Investigator and is found to be satisfactory. A lower dose may be chosen if deemed appropriate following review of PK and safety data from Part A.

Subjects will be admitted to the clinical unit in the morning of Day -1 and will remain in the unit until the scheduled assessments and procedures have been performed on Day 7, 48 h post-last dose. On Day -1 subjects' eligibility will be re-assessed and blood and urine samples will be collected for laboratory safety tests (including drugs of abuse and alcohol screen, biochemistry, haematology, urinalysis and serum pregnancy test). A 12-lead ECG, vital signs (supine systolic and diastolic blood pressure, pulse), body temperature, quantitative sensory testing (QST) and visual analogue scale (VAS) and adverse event and concomitant medication checks will be performed. The intravenous dose of BN201 or placebo will be based on body weight measured on Day -1. An evening snack will be consumed at least 10 h before (each) dose administration.

After an overnight fast of at least 10 h, dose administration will occur on the mornings of Day 1 to Day 5 between 08:00 and 11:00 whilst subjects are in a semi supine position. The subjects will remain in this position until 2 h post-infusion, however other positions are temporarily allowed for scheduled assessment requirements. Fasting will continue until 4 h after start of infusion; a standardised meal will then be administered.

Subjects will be discharged from the clinical unit on Day 7 providing there are no ongoing safety concerns. The following assessments will be made during Day -1 to Day 7:

* Safety assessments: Adverse event (AEs) and concomitant medication check, physical examination, laboratory safety assessments (drugs of abuse and alcohol screen, biochemistry, haematology and urinalysis and serum pregnancy test), 12-lead ECG, telemetry, Holter monitoring, EEG monitoring*, vital signs (supine systolic and diastolic blood pressure, pulse) and body temperature, infusion site reaction assessment, C-SSRS questionnaire, QST and VAS.
* PK assessments: Blood sample collection for measurement of BN201 in plasma.
* PD assessments: Blood sample collection for measurement of phosphorylation of N-myc downstream-regulated gene 1 (NDGR1) in peripheral blood mononuclear cells (PBMCs).
* Pharmacogenomic assessments: Blood sample will be collected for potential genotyping of deoxyribonucleic acid (DNA) sequence variants to explore potential relationships with PK/PD and or tolerability.

  * EEG monitoring only performed for Part B Cohort 2 if indicated from results from Part B Cohort 1

A follow-up visit (including a brain MRI scan) will be conducted 12 to 16 days following the subjects' final administration of IMP. If all follow up assessments are satisfactory to the Investigator, the subject will be discharged from the study. If any AEs are ongoing, or any assessments not satisfactory subjects may be recalled to the unit for follow-up assessments until the Investigator is satisfied the subject may be discharged from the study. Subjects will be advised to return or contact the unit at any time if they may be experiencing any adverse effects.

ELIGIBILITY:
Inclusion Criteria:

To be confirmed at screening:

1. Healthy male and female subjects between 18 and 55 years of age.
2. *Healthy subjects as determined by past medical history and as judged by the PI (including no significant infection in the last 3 months before trial enrolment).
3. *Female subject of non-child bearing potential with negative pregnancy test at screening and each admission to the clinical unit. For the purposes of this study, this is defined as the subject being amenorrheic for at least 12 consecutive months or at least 4 months post-surgical sterilisation (including bilateral fallopian tube ligation or bilateral oophorectomy with or without hysterectomy). Menopausal status will be confirmed by demonstrating at screening that levels of follicle stimulating hormone (FSH) fall within the respective pathology reference range. In the event a subject's menopause status has been clearly established (for example, the subject indicates she has been amenorrheic for 10 years), but FSH levels are not consistent with a post-menopausal condition, determination of subject eligibility will be at Investigator's discretion following consultation with the Sponsor.
4. *Female subjects of child bearing potential must be non-pregnant and non-lactating with negative pregnancy test at screening and each admission to the clinical unit.
5. *Female subjects of child bearing potential and male subjects with female partners of child bearing potential must take one highly effective contraceptive precaution in addition to one acceptable contraceptive precaution (i.e., barrier precaution) from first dose until 3 months after last dose of IMP (as detailed in Section 9.4.1).
6. *Male subject willing to use an effective method of contraception or 2 effective methods of contraception, i.e., highly effective method of contraception + condom, if applicable (unless anatomically sterile or where abstaining from sexual intercourse is in line with the preferred and usual lifestyle of the subject) from first dose until 3 months after last dose of IMP.
7. *Subject with a body weight of ≥ 50.0 kg and ≤100 kg and have a body mass index (BMI) of 18-32 kg/m2. BMI = body weight (kg) / [height (m)]2.
8. *Subject with no clinically significant history of previous allergy / sensitivity to BN201 or any of the excipients contained within the IMP.
9. *Subject with no clinically significant abnormal serum biochemistry, haematology and urine examination values within 28 days before the first dose of IMP.
10. *Subject with a negative urinary drugs of abuse screen, determined within 28 days before the first dose of IMP (N.B. a positive alcohol result may be repeated at Investigator's discretion).
11. Subject with negative human immunodeficiency virus (HIV) and hepatitis B surface antigen (HBsAg) and hepatitis C virus antibody (HCV) results.
12. *Subject with no clinically significant abnormalities in 12-lead electrocardiogram ((QTcF ≤ 430 ms) and (PR 120 - 200 ms)) determined within 28 days before first dose of IMP.
13. Subjects with no clinically significant abnormalities in electroencephalogram (EEG) determined within 28 days before first dose of IMP.
14. *Subject with no clinically significant abnormalities in vital signs (supine systolic and diastolic blood pressure, pulse) and body temperature determined within 28 days before first dose of IMP.
15. Subject must be available to complete the study (including all follow up visits).
16. Subject must satisfy the investigator / designee about their fitness to participate in the study.
17. Subject must be willing and able to sign the written informed consent to participate in the study.
18. Subjects must not donate sperm for the first dose and for at least 3 months after the last dose of IMP.
19. Subject with no clinically significant abnormalities in brain MRI scan determined within 28 days before first dose of IMP.

To be re-confirmed on Day -1 / prior to dosing:

1. Subject continues to meet all screening inclusion criteria indicated with * (BMI will only apply to screening).
2. Subject with a negative urinary drugs of abuse screen (including alcohol) prior to dosing.
3. Female subject with negative pregnancy test.

Exclusion Criteria:

To be confirmed at screening:

1. Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements within 14 days or 5 half-lives (whichever is longer) prior to the first dose of IMP, unless in the opinion of the Investigator the medication will not interfere with the study procedures or compromise subject safety.
2. Evidence of renal, hepatic, central nervous system, respiratory, cardiovascular or metabolic dysfunction.
3. A clinically significant history of drug or alcohol abuse.
4. Users of nicotine products i.e., current smokers or ex-smokers who have smoked within the 6 months prior to dosing with the study medication or users of cigarette replacements (i.e., e-cigarettes, nicotine patches or gums).
5. Inability to communicate well with Investigators (i.e., language problem, poor mental development or impaired cerebral function).
6. Participation in a New Chemical Entity clinical study within the previous 3 months or a marketed drug clinical study within the 30 days before the first dose of IMP. (Washout period between studies is defined as the period of time elapsed between the last dose of the previous study and the first dose of the next study).
7. Donation of 450 mL or more blood within the 3 months before the first dose of IMP.

To be re-confirmed at Day -1 / prior to dosing:

1. Development of any exclusion criteria since screening.
2. Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements since screening, unless in the opinion of the Investigator and Sponsor's Responsible Physician the medication will not interfere with the study procedures or compromise subject safety.
3. Participation in a clinical study since the screening visit.
4. Donation of 450 mL or more blood within the 3 months before the first dose of IMP and until at least 3 months after the final study visit.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2018-05-27 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-22 (Actual)

PRIMARY OUTCOMES:
Safety: Adverse Events (AEs) and serious adverse events (SAEs) Reporting | Up to 17 days
  All AEs will be recorded, whether considered minor or serious, drug-related or not.
Safety: Routine Laboratory Safety Screen on Haematology | Up to 17 days
  Analysis for Haematology
Safety: Routine Laboratory Safety Screen on Urinary Sodium | Up to 17 days
  Analysis for Urinary Sodium
Safety: Routine Laboratory Safety Screen on Biochemistry | Up to 17 days
  Analysis for Biochemistry
Safety: Routine Laboratory Safety Screen on Urinary Potassium | Up to 17 days
  Analysis for Urinary Potassium
Safety: Vital signs Measures on Systolic blood pressure | Up to 17 days
  Check of Systolic blood pressure
Safety: Vital signs Measures on Diastolic blood pressure | Up to 17 days
  Check of Diastolic blood pressure
Safety: Vital signs Measures on oral body temperature | Up to 17 days
  Check of oral body temperature
Safety: Vital signs Measures on Pulse rate | Up to 17 days
  Check of pulse rate
Magnetic resonance imaging (MRI) brain scan | Up to 17 days
  Non-contrast MRI brain scans
Safety: Suicide Risk assessement | Up to 17 days
  Assessment of Suicide-related thoughts and behaviours using Columbia-Suicide Severity Rating Scale (C-SSRS) Questionnaire
Safety: Physical Examination for ear | Up to 17 days
  Examination of ear
Safety: 12-lead Electrocardiography (ECG) Recording | Up to 17 days
  Performance of ECGs in the supine position
Safety: Telemetry Monitoring | Up to 5 days
  Cardiac rhythm measure
Safety: Pain report | Day 5
  Spontaneous (neuropathic) pain report using Visual Analogue Scale (VAS) tool
Safety: Quantitative Sensory Testing (QST) | Day 5
  Evaluation of increase in mechano-sensitivity
Safety: Infusion Site Reaction Assessment | Up to 17 days
  Assessment of Infusion Site Reaction
Safety: Holter Monitoring | Up to 5 days
  Cardiac rhythm measure
Safety: Electroencephalography (EEG) Recording | Up to 5 days
  Electrical activity measure
Safety: Concomitant Medication Recording | Up to 17 days
  All prior and concomitant medications taken record
Safety: Physical Examination for nose | Up to 17 days
  Examination of nose
Safety: Physical Examination for throat | Up to 17 days
  Examination of throat
Safety: Physical Examination for eye | Up to 17 days
  Examination of ophthalmological aspects
Safety: Physical Examination for skin | Up to 17 days
  Examination of dermatological aspects
Safety: Physical Examination for cardiovascular | Up to 17 days
  Examination of cardiovascular aspects
Safety: Physical Examination for Respiratory | Up to 17 days
  Examination of respiratory aspects
Safety: Physical Examination for gastrointestinal | Up to 17 days
  Examination of gastrointestinal aspects
Safety: Physical Examination for Central Nervous System | Up to 17 days
  Examination of central nervous system
Safety: Physical Examination for Lymph Nodes | Up to 17 days
  Examination of lymph nodes
Safety: Physical Examination for musculoskeletal | Up to 17 days
  Examination of musculoskeletal aspects

SECONDARY OUTCOMES:
Pharmacokinetic Parameter: Cmax measurement | From pre-dose to 24 hours post-start-infusion
  Maximum concentration measurement in plasma
Pharmacokinetic Parameter: Tm concentration measurement | From pre-dose to 24 hours post-start-infusion
  Time to maximum observed concentration in plasma
Pharmacokinetic Parameter: kel measurement | From pre-dose to 24 hours post-start-infusion
  Elimination rate constant in plasma
Pharmacokinetic Parameter: t1/2 measurement | From pre-dose to 24 hours post-start-infusion
  Terminal elimination half-life in plasma
Pharmacokinetic Parameter: AUC 0-τ measurement | From pre-dose to 24 hours post-start-infusion
  Area under the concentration-time curve (AUC) from 0 to τ, where τ is the dosing interval (0 - 24 h) in plasma
Pharmacokinetic Parameter: AUC 0-t measurement | From pre-dose to 24 hours post-start-infusion
  Area under the concentration-time curve (AUC) from the time of dosing to the time of the last measurable concentration in plasma
Pharmacokinetic Parameter: AUC 0-inf measurement | From pre-dose to 24 hours post-start-infusion
  AUC extrapolated to infinity
Pharmacokinetic Parameter: AUC % measurement | From pre-dose to 24 hours post-start-infusion
  extrapolated Residual area
Pharmacokinetic Parameter: Clearance (CL) measurement | From pre-dose to 24 hours post-start-infusion
  Clearance
Pharmacokinetic Parameter: Vz measurement | From pre-dose to 24 hours post-start-infusion
  Volume of distribution

OTHER OUTCOMES:
Pharmacodynamic Parameter: Phosphorylation of N-myc downstream regulated 1 (NDRG1) measurement | Up to 2 hours post start infusion
  NDRG1 phosphorylation in PBMCs
Pharmacogenomics Parameter: Sequencing of DNA in blood samples | Day 1
  Potential genotyping of deoxyribonucleic acid (DNA) sequence variants in blood sample

CONTACTS AND LOCATIONS:
Overall Officials: Annelize Koch, MBChB, Principal Investigator — Simbec Research
Locations (1):
- Simbec Research Limited, Merthyr Tydfil, United Kingdom

IPD SHARING:
Plan to Share IPD: No